CLINICAL TRIAL: NCT03075332
Title: Detraining in the Components of Physical Aptitude in People Living With HIV/ AIDS
Brief Title: Detraining in People Living With HIV/AIDS
Acronym: PVHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, JULIANY DE SOUZA ARAUJO, principal investigator, Universidade Federal do Rio Grande do Norte
Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VIVER MAIS
Record Dates: First submitted 2017-02-09; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-02

CONDITIONS: Lipodystrophy Syndrome, HIV; Sarcopenia
Keywords: Detraining; Physical aptitude; HIV
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; Sarcopenia

STUDY DESIGN:
Intervention Model Description: This is a longitudinal study of the non-randomized experimental type, presenting a non-probabilistic sample for convenience and independent groups. The sample consisted of 21 individuals divided into 2 groups: Experimental Group (EG) and Control Group (CG). The EG was composed of 11 people living with HIV/AIDS and CG composed of 10 people with no infection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- protocol with physical exercise (Experimental): Both groups underwent a combined training intervention consisting of aerobic and resisted exercises in the same training session
  Interventions: Other: combined training

INTERVENTIONS:
Other: combined training — Combined training consisting of aerobic and resisted training in the same training session for 15 weeks followed by 5 weeks of detraining

SUMMARY:
The goal of this study was to evaluate the effect of detraining in the components of physical aptitude of people living with HIV/Aids (PVHA).

DETAILED DESCRIPTION:
The study was experimental with a sample composed by an Experimental Group (EG) with 11 PVHA, under antiretroviral therapy and a Control Group (CG) with 10 individuals without the infection; all which were under medical release and insufficiently active. The body composition was evaluated through the DXA, as well as the cardiorespiratory aptitude through the ergometer and the strength of the upper and lower limbs through dynamometry. Both groups conducted interventions with concurrent training for 15 weeks and the interruption of exercise was evaluated after a period of 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Group experience to have a diagnosis of at least 2 years living with HIV / AIDS being in clinical follow-up in the Specialized Attention Services in HIV / AIDS (SAE), using ART, TCD4 lymphocyte count equal to or greater than 500 copies / mm³, viral load Undetectable (≤ 50 copies / mm³)
* Group control without any diagnosis of HIV / AIDS or any other pathology. Both groups completed the exercise program with a minimum frequency of 75%.

Exclusion Criteria:

* Both groups taking part in any physical exercise in time of detraining

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2016-06-21 (Actual); Study Completion 2016-07-23 (Actual)

PRIMARY OUTCOMES:
Capacity cardiorespiratory | 21 weeks
  ml (cardiorespiratory aptitude through the ergometer)

SECONDARY OUTCOMES:
test force | 21 weeks
  kg (strength of the upper and lower limbs through dynamometry)

OTHER OUTCOMES:
body composition | 21 weeks
  kg (body composition was evaluated through the DXA)

CONTACTS AND LOCATIONS:
Overall Officials: juliany araujo, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (2):
- Brazil (2):
  - Juliany de Souza Araujo, Natal, Rio Grande do Norte
  - Juliany de Souza Araujo, Parnamirim, Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: Undecided
It is not done sharing since the individuals involved in the people are vulnerable and the secrecy is rescued

REFERENCES:
- [Background] Warshaw MG, Carey VJ, McFarland EJ, Dawson L, Abrams E, Melvin A, Fairlie L, Spiegel H, Jay J, Agwu AL; IMPAACT P1094 Team. The interaction between equipoise and logistics in clinical trials: A case study. Clin Trials. 2017 Jun;14(3):314-318. doi: 10.1177/1740774517690734. Epub 2017 Jan 31. PMID 28135804
- [Background] Li A, McCabe T, Silverstein E, Dragan S, Salbach NM, Zobeiry M, Beldick S, Godi C, O'Brien KK. Community-Based Exercise in the Context of HIV: Factors to Consider when Developing and Implementing Community-Based Exercise Programs for People Living with HIV. J Int Assoc Provid AIDS Care. 2017 May/Jun;16(3):267-275. doi: 10.1177/2325957416686836. Epub 2017 Jan 11. PMID 28074681
- [Background] Gomes Neto M, Conceicao CS, Oliveira Carvalho V, Brites C. Effects of Combined Aerobic and Resistance Exercise on Exercise Capacity, Muscle Strength and Quality of Life in HIV-Infected Patients: A Systematic Review and Meta-Analysis. PLoS One. 2015 Sep 17;10(9):e0138066. doi: 10.1371/journal.pone.0138066. eCollection 2015. PMID 26378794
- [Background] Poton R, Polito M, Farinatti P. Effects of resistance training in HIV-infected patients: A meta-analysis of randomised controlled trials. J Sports Sci. 2017 Dec;35(24):2380-2389. doi: 10.1080/02640414.2016.1267389. Epub 2016 Dec 21. PMID 28001474
- [Background] Chitu-Tisu CE, Barbu EC, Lazar M, Bojinca M, Tudor AM, Hristea A, Abagiu AO, Ion DA, Badarau AI. Body composition in HIV-infected patients receiving highly active antiretroviral therapy. Acta Clin Belg. 2017 Feb;72(1):55-62. doi: 10.1080/17843286.2016.1240426. Epub 2016 Oct 11. PMID 27724840
- [Derived] Araujo JS, de Medeiros RCDSC, da Silva TAL, de Medeiros DC, de Medeiros JA, Dos Santos IK, Wilde P, Cabral BGAT, Medeiros RMV, Dantas PMS. Effect of Training and Detraining in the Components of Physical Fitness in People Living With HIV/AIDS. Front Physiol. 2021 Sep 22;12:586753. doi: 10.3389/fphys.2021.586753. eCollection 2021. PMID 34630129
- Available data/document: Ethics committee project: plataforma brasil — http://aplicacao.saude.gov.br/plataformabrasil/visao/pesquisador/gerirPesquisa/gerirPesquisaAgrupador.jsf — all project